CLINICAL TRIAL: NCT00227123
Title: A Randomized Control Trial Comparing Quetiapine to Risperidone in Bipolar Disorder Outpatients With Current Stimulant Dependence
Brief Title: A Randomized Control Trial Comparing Quetiapine to Risperidone in Bipolar Disorder With Stimulant Dependence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Stanley Medical Research Institute (Other); University of North Texas Health Science Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0602342; 02T147
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Last update posted 2008-01-04 (Estimated); Status verified 2007-10

CONDITIONS: Bipolar Disorder; Cocaine Dependence; Methamphetamine Dependence
Keywords: Bipolar, cocaine, methamphetamine,quetiapine,risperidone
MeSH Terms: conditions — Bipolar Disorder; Cocaine-Related Disorders | interventions — Quetiapine Fumarate; Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator): Quetiapine versus Risperidone
  Interventions: Drug: quetiapine, risperidone

INTERVENTIONS:
Drug: quetiapine, risperidone — Flexible dose titrations to 'treat-to-symptoms'
  Other Names: Seroquel; Risperdal

SUMMARY:
The purpose of this study is to determine whether quetiapine or risperidone are effective in treating mood symptoms, drug cravings and use in bipolar disorder with concurrent cocaine or methamphetamine dependence.

DETAILED DESCRIPTION:
Bipolar disorder may be associated with the highest rates of substance abuse of any psychiatric illness. Studies suggest that substance abuse in persons with bipolar disorder have lifetime prevalence rates as high as 60% with reports of cocaine abuse as high as 30%. Comorbid substance abuse in persons with bipolar disorder is associated with increased hospitalization, poorer psychiatric recovery and treatment response than in patients with bipolar disorder alone. Thus, therapeutic agents that may enhance prognosis by improving psychiatric outcomes, reducing stimulant cravings, and increasing treatment retention are of considerable interest. In a previous study conducted in this lab, we found that conventional neuroleptic agents were associated with an increase in depressive symptoms and a significant increase in stimulant cravings. These results mirror preclinical animal data that show conventional neuroleptics (i.e.haloperidol) with high dopamine receptor binding affinities actually increase cocaine self-administration in rats and monkeys. These results are clinically relevant as persons with bipolar disorder who abuse cocaine and other drugs often receive higher doses of conventional neuroleptics than those without cocaine or other drug abuse. In contrast to conventional neuroleptic therapy, atypical antipsychotics (i.e. quetiapine, risperidone), decrease self-administration of cocaine. The receptor binding profile of the atypical antipsychotics broadly vary although all agents in this drug class are known as serotonin-dopamine antagonists. Quetiapine has 'moderate' dopamine binding, while risperidone has 'high' dopamine receptor binding properties similar to conventional neuroleptic agents. Thus, our hypothesis is that quetiapine may be a more efficacious agent than risperidone in treating bipolar mood symptoms while attenuating drug cravings and use.

ELIGIBILITY:
Inclusion criteria:

1. English-speaking men and women (20-50 years old) of all ethnic origins
2. Outpatients with a current DSM-IV diagnosis of bipolar I with or without psychotic features or bipolar II disorder
3. Current cocaine or methamphetamine dependence
4. Currently experiencing hypomanic, manic, or mixed state episodes with a Young Mania Rating Scale23 (YMRS11) score of > 9
5. Currently craving stimulants with a craving score of > 20 on the 10-item, self-reported Stimulant Craving Questionnaire24 (SCQ10)
6. A high school diploma, GED, or Shipley IQ test score of >85.

Exclusion criteria:

1. Inpatients or anyone with a high risk for suicide (i.e., active suicidal ideation with a proposed plan, history of any suicide attempt within the last 6 months)
2. DSM-IV diagnosis of substance-induced mood disorder
3. Pregnant or breast-feeding
4. History of special education, mental retardation, dementia
5. HIV/AIDS, reactive hepatitis, hepatic cirrhosis or any active liver disease, personal or familial history of diabetes, personal history of heart disease (i.e., congenital heart abnormalities, congestive heart failure, chronic atrial fibrillation, rheumatic heart disease, heart attack)
6. Central nervous system diseases (e.g., multiple sclerosis, severe head trauma, or seizures)
7. Contraindications or allergic reactions to study medications
8. Currently participating in any other research program
9. Urine positive for glucose or ketones
10. Currently receiving any antipsychotic medications or more than two psychotropic medications
11. Currently receiving benzodiazepines, sedatives or stimulants
12. Any other current substance dependence
13. Cataracts or glaucoma
14. EKG evidence of QT prolongation.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2002-10; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Mood symptom improvement. | Baseline to exit
Cocaine or methamphetamine cravings and use. | Baseline to exit

SECONDARY OUTCOMES:
Body Mass Index | Baseline to Exit

CONTACTS AND LOCATIONS:
Overall Officials: Vicki A. Nejtek, Ph.D., Principal Investigator — University of North Texas Health Science Center
Locations (2):
- United States (2):
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Universty of North Texas Health Science Center, Fort Worth, Texas

REFERENCES:
- [Derived] Nejtek VA, Avila M, Chen LA, Zielinski T, Djokovic M, Podawiltz A, Kaiser K, Bae S, Rush AJ. Do atypical antipsychotics effectively treat co-occurring bipolar disorder and stimulant dependence? A randomized, double-blind trial. J Clin Psychiatry. 2008 Aug;69(8):1257-66. doi: 10.4088/jcp.v69n0808. PMID 18681757